CLINICAL TRIAL: NCT02341716
Title: Hospital- or Home-based Supervised Exercise Therapy or Unsupervised Walk Advice for Patients With Intermittent Claudication
Brief Title: Hospital- and Home-based Supervised Exercise Versus UNsupervised Walk Advice For Patients With InTermittent Claudication
Acronym: SUNFIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lennart Jivegård (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor-Investigator, Lennart Jivegård, MD, University lecturer, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SahlgrenskaUH
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Intermittent Claudication
Keywords: intermittent claudication; exercise therapy; physiotherapy
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Walk advice (Active Comparator): All WA patients receive best medical treatment (BMT) including control of risk factors for arteriosclerosis, simvastatin 40 mg daily, aspirin 75 mg daily and are recommended outdoor walking with Nordic Poles at least 30 minutes at least three times per week. The WA patients are unsupervised during the study period and are followed by a blinded observer at baseline, three, six and 12 months.
  Interventions: Procedure: WA
- Hospital-based supervised exercise (Active Comparator): All SET patients receive the same basic treatment as WA patients: best medical treatment (BMT) including control of risk factors for arteriosclerosis, simvastatin 40 mg daily, aspirin 75 mg daily and recommendation of outdoor walking with Nordic Poles at least 30 minutes at least three times per week. The SET group in addition receives three times weekly during six months in-hospital muscle exercise therapy in a group supervised by a physiotherapist. After the six months of supervised exercise therapy, the SET patients are recommended to continue the same muscle exercise therapy at home, but without feedback, between seven and 12 months.
  Interventions: Procedure: SET
- Home-based supervised exercise (Active Comparator): All HET patients receive the same basic treatment as WA patients: best medical treatment (BMT) including control of risk factors for arteriosclerosis, simvastatin 40 mg daily, aspirin 75 mg daily and recommendation of outdoor walking with Nordic Poles at least 30 minutes at least three times per week. The HET group patients in addition perform the same muscle exercise therapy three times weekly during six months as the SET patients, but in their homes, and are supervised and given feedback by phone calls every 14th day by a physiotherapist. After six months of supervised exercise therapy, the HET patients are recommended to continue the same muscle exercise therapy, but without feedback, between seven and 12 months.
  Interventions: Procedure: HET

INTERVENTIONS:
Procedure: WA — Walk advice with Nordic Poles and best medical treatment
  Arms: Walk advice
Procedure: SET — Walk advice with Nordic Poles, best medical treatment and hospital-based supervised exercise therapy
  Arms: Hospital-based supervised exercise
Procedure: HET — Walk advice with Nordic Poles, best medical treatment and home-based supervised exercise therapy
  Arms: Home-based supervised exercise

SUMMARY:
The purpose of this randomized clinical trial is to determine and compare the clinical and cost effectiveness of three methods for exercise therapy as treatment for patients with intermittent claudication. The methods tested are a hospital-based (SET) and a home-based (HET) supervised exercise program and unsupervised walk advice (WA) and all patients are followed for 12 months. Unsupervised WA consists of advice of at least 30 minutes walking with Nordic Poles (NP) at least three times per week and this basic treatment, including best medical treatment, is used in all three treatment groups. In addition to this basic treatment, the SET group patients during the first six months participate in group-based exercise therapy in the hospital for 50 minutes three times weekly, supervised by a physiotherapist. The HET group patients perform the same exercise in their home 50 minutes three times weekly during six months receiving feedback from a physiotherapist by a phone call every 14th day. The SET and HET group patients are recommended to continue the 50 minutes three times weekly exercise therapy in their homes without supervision during the last six months. Primary outcome is change from baseline to 12 months in walking distance during six minutes in a hospital corridor (6MWT) and co-primary outcome is change from baseline to 12 months in health-related quality of life (HRQoL) using the SF36 questionnaire. Secondary outcomes include fulfillment of patient-specified goals with treatment (PSFS), change in health-related quality-of-life (HRQoL) with a disease-specific instrument (VascuQoL), walking impairment as measured by the Walking Impairment Questionnaire, physical activity (accelerometer) and compliance with physical exercise therapy (patient diary).

DETAILED DESCRIPTION:
Background Intermittent claudication is usually caused by atherosclerotic stenoses and/or occlusions in the arteries to the legs and affects 7% of the Swedish population aged 60 years or more. Evidence-based treatment is best medical treatment (BMT) and exercise therapy. Best medical treatment includes treatment of risk factors for arteriosclerosis. Regarding exercise therapy, in-hospital supervised exercise therapy (SET) on a graded treadmill is known to improve walking performance as measured on the graded treadmill after three and six months. There is only scarce data on long-term results and very limited data regarding improvement of health related quality of life (HRQoL) by SET. In most countries, walk advice (WA) is routine clinical practice and resources for SET are often lacking. Invasive treatment (surgical or endovascular) is rarely required for patients with intermittent claudication.

New techniques (GPS and accelerometers) enable measurement of physical activity and training in home environment. The use of such techniques could facilitate home-based (HET) instead of hospital-based supervised exercise (SET) therapy by providing the caregiver data that could be used for feedback to the patient in order to obtain optimal patient benefit by the exercise therapy. This raises hope that results of and the long-term compliance to exercise therapy may improve.

Aim: in patients with intermittent claudication (IC) who do not require invasive treatment evaluate walking performance, HRQoL, fulfillment of patient-defined goals with treatment, walking impairment, long-term compliance to exercise therapy, physical activity and cost-effectiveness for different exercise therapy modalities in order to define the most effective and cost effective treatment.

One hundred and sixty-five IC patients requesting treatment for their IC symptoms in the vascular surgical departments of Sahlgrenska University Hospital and Södra Älvsborg Hospital, Sweden and in whom invasive treatment is not considered necessary are randomized (computerized adaptive stratified randomization) to

1. WA with Nordic Poles (NP) + best medical treatment (BMT), or
2. WA with NP + BMT + SET, or
3. WA with NP + BMT + HET

All randomized patients are recommended outdoor walking with NP at least 30 minutes at least three times per week. The SET group in addition receives in-hospital muscle exercise therapy in a group supervised by a physiotherapist three times weekly during six months. The HET group patients perform the same muscle exercise therapy at home with feedback every 14th day from a physiotherapist during six months. After the six months of supervised exercise therapy, the SET and HET patients are recommended to continue the same muscle exercise therapy at home, but without feedback, between seven and 12 months. The patients are followed by a blinded observer (physiotherapist unaware of the patient´s randomized group) at three, six and 12 months.

Primary outcome: change from baseline to 12 months in walking distance during six-minutes-walk-test (6MWT) and co-primary outcome: change from baseline to 12 months in health-related quality of life (SF36).

Secondary outcomes: walking impairment as measured by the Walking Impairment Questionnaire (WIQ), fulfillment of patient-defined goals (Patient-Specific-Functional Scale), physical activity (accelerometer), compliance to exercise therapy (patient diary), disease-specific HRQoL (VascuQol) and cost-effectiveness. Also change over time (baseline to three, baseline to six and six to 12 months) is studied.

It is important to determine whether the supervised exercise therapy modalities (SET and HET) have equivalent results and are better than WA with NP and BMT alone. The trial is designed to answer the question whether HET is not significantly less clinically effective as SET and whether SET is more clinically effective than WA with NP and BMT. The study started in September 2014, inclusion is expected to stop in September 2016 and end of follow-up is September 2017.

ELIGIBILITY:
Inclusion Criteria:

1. Intermittent claudication in one or both legs with a typical history and ankle-brachial-index (ABI) 0.90 or less and/or 30% or more post-exercise reduction of ABI.
2. Symptom duration > 6 months.
3. Intermittent claudication is the walk limiting condition.

Exclusion Criteria:

1. Invasive treatment for intermittent claudication performed within three months
2. Invasive treatment for intermittent claudication considered necessary within 12 months
3. Inability to understand Swedish, answer questionnaires or perform walk test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Six-minutes-walk-test walking distance (6MWD) | Baseline and 12 months, change
  Walk test in a hospital corridor where the patient is encouraged to walk as far as possible between two cones, 30 meters apart, during six minutes
Generic health-related quality of life (SF36) | Baseline and 12 months, change
  Short-form 36 is an extensively used and validated generic health-related quality of life instrument

SECONDARY OUTCOMES:
Disease-specific health-related quality of life (VascuQoL) | Baseline and 12 months, change
  VascuQoL is a frequently used disease-specific (PAD) HRQoL instrument, validated in Swedish.
Walking impairment (Walking Impairment Questionnaire, WIQ) | Baseline and 12 months, change
  The WIQ questionnaire is a frequently used questionnaire to quantify walking impairment and is validated in Swedish
Physical activity | Baseline and 12 months, change
  Physical activity is assessed using an accelerometer (ActivePAL) carried by the patient during one week adhered to the thigh and covered with a plastic foil to allow a shower. The ActivePAL gives continuous data (e.g. standing, sitting, walking) regarding physical activity and is validated for use in patients with intermittent claudication
Compliance to exercise therapy | 12 months
  Compliance to exercise therapy is assessed by a patient diary in which the patients register all exercise activities (SET and HET groups only)
HbA1c and serum lipids | Baseline and 12 months, change
  Standard blood tests
Ankle-brachial-index (ABI) | Baseline and 12 months, change
  The highest pressure at the ipsilateral ankle level divided by the simultaneously measured arm blood pressure
Patient-specified goals with treatment (PSFS) | 12 months
  At baseline, the patient specifies one to five goals with the treatment for intermittent claudication and fulfillment of these goals is quantified by the patient during follow-up
Cardiovascular events | 12 months
  Cardiovascular adverse events, minor and major, during the course of the study
Muscular-skeletal events | 12 months
  Muscular-skeletal events, minor and major, during the course of the study
Vascular surgical revascularization | 12 months
  Invasive vascular procedure in the lower limb(s) during the course of the study
Six-minutes-walk-test walking distance (6MWD) | Baseline and three months, change
  Walk test in a hospital corridor where the patient is encouraged to walk as far as possible between two cones, 30 meters apart, during six minutes
Six-minutes-walk-test walking distance (6MWD) | Baseline and six months, change
  Walk test in a hospital corridor where the patient is encouraged to walk as far as possible between two cones, 30 meters apart, during six minutes
Six-minutes-walk-test walking distance (6MWD) | Six and 12 months, change
  Walk test in a hospital corridor where the patient is encouraged to walk as far as possible between two cones, 30 meters apart, during six minutes
Generic health-related quality of life (SF36) | Baseline and three months, change
  Short-form 36 is an extensively used and validated generic health-related quality of life instrument
Generic health-related quality of life (SF36) | Baseline and six months, change
  Short-form 36 is an extensively used and validated generic health-related quality of life instrument
Generic health-related quality of life (SF36) | Six and 12 months, change
  Short-form 36 is an extensively used and validated generic health-related quality of life instrument
Disease-specific health-related quality of life (VascuQoL) | Baseline and three months, change
  VascuQoL is a frequently used disease-specific (PAD) HRQoL instrument, validated in Swedish.
Disease-specific health-related quality of life (VascuQoL) | Baseline and six months, change
  VascuQoL is a frequently used disease-specific (PAD) HRQoL instrument, validated in Swedish.
Disease-specific health-related quality of life (VascuQoL) | Six and 12 months, change
  VascuQoL is a frequently used disease-specific (PAD) HRQoL instrument, validated in Swedish.
Walking impairment (Walking Impairment Questionnaire, WIQ) | Baseline and three months, change
  The WIQ questionnaire is a frequently used questionnaire to quantify walking impairment and is validated in Swedish
Walking impairment (Walking Impairment Questionnaire, WIQ) | Baseline and six months, change
  The WIQ questionnaire is a frequently used questionnaire to quantify walking impairment and is validated in Swedish
Walking impairment (Walking Impairment Questionnaire, WIQ) | Six and 12 months, change
  The WIQ questionnaire is a frequently used questionnaire to quantify walking impairment and is validated in Swedish
Physical activity | Baseline and three months, change
  Physical activity is assessed using an accelerometer (ActivePAL) carried by the patient during one week adhered to the thigh and covered with a plastic foil to allow a shower. The ActivePAL gives continuous data (e.g. standing, sitting, walking) regarding physical activity and is validated for use in patients with intermittent claudication
Physical activity | Baseline and six months, change
  Physical activity is assessed using an accelerometer (ActivePAL) carried by the patient during one week adhered to the thigh and covered with a plastic foil to allow a shower. The ActivePAL gives continuous data (e.g. standing, sitting, walking) regarding physical activity and is validated for use in patients with intermittent claudication
Physical activity | Six and 12 months, change
  Physical activity is assessed using an accelerometer (ActivePAL) carried by the patient during one week adhered to the thigh and covered with a plastic foil to allow a shower. The ActivePAL gives continuous data (e.g. standing, sitting, walking) regarding physical activity and is validated for use in patients with intermittent claudication
Compliance to exercise therapy | Three months
  Compliance to exercise therapy is assessed by a patient diary in which the patients register all exercise activities (SET and HET groups only)
Compliance to exercise therapy | Six months
  Compliance to exercise therapy is assessed by a patient diary in which the patients register all exercise activities (SET and HET groups only)
Patient-specified goals with treatment (PSFS) | Six months
  At baseline, the patient specifies one to five goals with the treatment for intermittent claudication and fulfillment of these goals is quantified by the patient during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Jivegård, MD, Lecturer, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Södra Älvsborgs Hospital, Borås, Västra Götaland County
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County

REFERENCES:
- [Derived] Sandberg A, Back M, Cider A, Jivegard L, Sigvant B, Nordanstig J. Impact of walk advice alone or in combination with supervised or home-based structured exercise on patient-reported physical function and generic and disease-specific health related quality of life in patients with intermittent claudication, a secondary analysis in a randomized clinical trial. Health Qual Life Outcomes. 2023 Oct 23;21(1):114. doi: 10.1186/s12955-023-02198-8. PMID 37872617
- [Derived] Sandberg A, Nordanstig J, Cider A, Jivegard L, Hagstromer M, Back M. The Impact of Nordic Pole Walk Advice Alone or in Combination With Exercise Strategies on Daily Physical Activity in Patients With Intermittent Claudication: A Randomized Clinical Trial. Phys Ther. 2023 Nov 4;103(11):pzad086. doi: 10.1093/ptj/pzad086. PMID 37459237
- [Derived] Sandberg A, Back M, Cider A, Jivegard L, Sigvant B, Wittboldt S, Nordanstig J. Effectiveness of supervised exercise, home-based exercise, or walk advice strategies on walking performance and muscle endurance in patients with intermittent claudication (SUNFIT trial): a randomized clinical trial. Eur J Cardiovasc Nurs. 2023 May 25;22(4):400-411. doi: 10.1093/eurjcn/zvac070. PMID 35917174
- [Derived] Sandberg A, Cider A, Jivegard L, Nordanstig J, Wittboldt S, Back M. Test-retest reliability, agreement, and minimal detectable change in the 6-minute walk test in patients with intermittent claudication. J Vasc Surg. 2020 Jan;71(1):197-203. doi: 10.1016/j.jvs.2019.02.056. Epub 2019 May 27. PMID 31147129